CLINICAL TRIAL: NCT00578851
Title: Post Approval Study of the C2a-Taper™ Acetabular System
Brief Title: A Clinical Investigation of the C2a-Taper™ Acetabular System
Status: Completed | Type: Observational
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: ORTHO.CR.H021; P050009 (Other: FDA)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Avascular Necrosis; Congenital Hip Dysplasia; Traumatic Arthritis
Keywords: Hip Arthroplasty; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- C2a Taper recipients: Patients who receive a THA with the C2a - Taper™ Acetabular System
  Interventions: Device: C2a - Taper™ Acetabular System

INTERVENTIONS:
Device: C2a - Taper™ Acetabular System — The C2a-Taper™ Acetabular System is a ceramic on ceramic hip articulating system. The bearing surfaces consist of ceramic femoral heads and acetabular liners.

SUMMARY:
The objective of this study is to gather clinical and survivorship information for the C2a-Taper™ Acetabular System, a ceramic-on-ceramic hip articulating system.

DETAILED DESCRIPTION:
Study Design:

Phase 1

Sites will collect the following types of data:

Clinical-Total Harris Hip Score, Radiographic Evaluation- measurements on acetabular and femoral components Survivorship-removal/revision of one or more components (i.e. liner, head, shell and/or stem) Safety- All other adverse events

Follow-up Visit schedule

* 6 week ± 2 weeks
* 6 month ± 1 month
* 1 year ± 3 months
* 2 years ± 3 months
* 3 years ± 3 months
* 4 years ± 3 months
* 5 years ± 3 months

Phase 2:

Patients continue to be followed on an annual basis (Years 6-10) via mail. A self assessment form is sent directly to the subject on an annual basis starting in the 6th post-operative year.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients with non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis, congenital hip dysplasia, and traumatic arthritis

Exclusion Criteria:

* Patients with: Osteoporosis, metabolic disorders, osteomalacia, rapid joint destruction, vascular insufficiency, muscular atrophy, and neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multi-Center study conducted in the United states on patients who meed the inclusion / exclusion criteria identified in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2006-04; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score, Radiographic Evaluation | 5 years

SECONDARY OUTCOMES:
Survivorship | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Zimmer Biomet
Locations (2):
- United States (2):
  - Physician's Clinic of Iowa, PCI, Cedar Rapids, Iowa
  - Lexington Clinic, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No